CLINICAL TRIAL: NCT07298928
Title: The Children's Hospital, Zhejiang University School of Medicine, National Clinical Research Center for Child Health
Brief Title: A Study on the Efficacy and Safety of Telitacicept in the Treatment of Children Ocular Myasthenia Gravis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Shanshan Mao, Directo, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYYS-2025-0347
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Effectiveness
Keywords: long-term follow-up; Ocular myasthenia gravis; Telitacicept; Children; Biological agent; Targeted treatment
MeSH Terms: conditions — Myasthenia Gravis | interventions — telitacicept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- a single Telitacicept treatment group (Experimental)
  Interventions: Drug: Telitacicept

INTERVENTIONS:
Drug: Telitacicept — All enrolled pediatric patients with OMG who meet the inclusion criteria will receive subcutaneous injections of Telitacicept on top of their existing medication regimen. The dose will be adjusted according to the patient's body weight: 160 mg per dose for those weighing ≥40 kg; 80 mg per dose for those weighing between 20 kg and <40 kg; for patients weighing <20 kg or aged <5 years, a gradual dose reduction may be considered based on individual circumstances. The administration schedule for Telitacicept (80 mg or 160 mg per dose) is as follows: once weekly via subcutaneous injection for the first 12 weeks; subsequently, once every two weeks via subcutaneous injection for the next 12 weeks; followed by once every four weeks via subcutaneous injection thereafter. Corticosteroids will be gradually tapered and discontinued based on changes in the patient's clinical condition.

SUMMARY:
Under conventional treatment regimens, pediatric ocular myasthenia gravis (OMG) is prone to relapse and is associated with corticosteroid-related adverse effects, indicating an unmet clinical need. In May 2025, the targeted B-cell biologic agent Telitacicept was approved for use in adult patients with acetylcholine receptor (AChR) antibody-positive generalized myasthenia gravis (GMG) and subsequently initiated in national multicenter clinical trials for adult OMG. Our center published a retrospective study in the Chinese Journal of Evidence-Based Pediatrics in August 2025, which was the first report both domestically and internationally on the efficacy and safety of Telitacicept in four pediatric OMG patients. This study plans to conduct a prospective, multicenter, open-label, single-arm clinical trial aimed at evaluating the effectiveness and safety of Telitacicept in pediatric OMG.

ELIGIBILITY:
Inclusion Criteria:

1. The patient and their legal guardian voluntarily sign the informed consent form.
2. Age < 18 years, male or female.
3. Diagnosis of OMG according to the Chinese Guidelines for the Diagnosis and Treatment of Myasthenia Gravis (2025 Edition).
4. Receiving corticosteroid therapy prior to enrollment.

Exclusion Criteria:

1. Active infection under treatment： Patients who are HBsAg positive must be excluded. Patients who are HBsAg negative but HBcAb positive must undergo quantitative HBV-DNA testing. Patients with a positive quantitative HBV-DNA result must be excluded; those with a negative result may be enrolled.
2. Severe hepatic or renal insufficiency.
3. Patients with malignant tumors other than thymoma.
4. Patients within 3 months post-thymectomy.
5. Hypogammaglobulinemia (IgG < 400 mg/dL) or IgA deficiency (IgA < 10 mg/dL).
6. History of allergy to human-derived biological products.
7. Participation in any other clinical trial within 28 days prior to enrollment or within 5 times the half-life of the investigational drug from the previous trial (whichever is longer).
8. Patients deemed unsuitable for participation by the investigator (e.g., patients with severe psychiatric disorders).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Ocular Myasthenia Gravis Rating Scale-q Score | baseline, 1 week, 2 week,3 week,4 week,6 week, 8 week, 10 week,12week, 16 week, 20 week, 24 week, 28 week, 32 week, 36 week, 40 week, 44 week, 48 week
  This Ocular Myasthenia Gravis Rating Scale (OMGRate) is used to assess the impact of symptoms on the quality of daily life in patients with OMG. The OMGRate-q section of the scale is the patient - reported outcome component for evaluating the improvement of self - perceived symptoms. The questionnaire is completed based on the patient's condition over the past 2 weeks.
  The total score ranges from 0 to 52 points, with higher scores indicating more severe symptoms and greater impairment of daily quality of life.

SECONDARY OUTCOMES:
quantitative Myasthenia Gravis scale | baseline, 1 week, 2 week,3 week,4 week,6 week, 8 week, 10 week,12week, 16 week, 20 week, 24 week, 28 week, 32 week, 36 week, 40 week, 44 week, 48 week
  This scale is a standardized tool for the objective measurement of muscle strength and endurance in MG-affected muscle groups. It consists of 13 items covering the following aspects: eyes (onset time of diplopia and ptosis), facial muscles (lip closure strength), pharynx and larynx (swallowing and pronunciation tests), respiration (percentage of forced vital capacity relative to the predicted value), neck (duration of head lifting while lying supine), hand strength (strength reduction measured by a dynamometer), and limbs (duration of posture maintenance).
  Each item is scored on a 4-point scale: 0 (normal), 1 (mild), 2 (moderate), and 3 (severe), with a total score ranging from 0 to 39. Higher scores indicate more severe symptoms.
Myasthenia Gravis⁃activity of daily living scale | baseline, 1 week, 2 week,3 week,4 week,6 week, 8 week, 10 week,12week, 16 week, 20 week, 24 week, 28 week, 32 week, 36 week, 40 week, 44 week, 48 week
  This scale is mainly used to assess the impact of symptoms on the quality of daily life in patients with MG and reflect the severity of the disease.
  It includes 8 items covering 4 aspects: eyes (frequency of ptosis and diplopia), bulbar region (degree of involvement in speech, chewing, and swallowing), respiration (relationship between breathing and physical activity), and limbs (ability to complete daily movements).
  Each item is scored on a scale of 0 (normal) to 3 (most severe), with a total score ranging from 0 to 24. Higher scores indicate greater disease severity.
The proportion of children patients who have their hormone therapy discontinued | 12week, 48 week

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Shenzhen children's Hospital of China Medical University, Shenzhen, Guangdong
  - Children's Hospital Affiliated to Shandong University, Jinan, Shandong
  - The Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No